CLINICAL TRIAL: NCT02137603
Title: Fast Track Appendectomy in Pediatric Patients With Intraoperative Findings of Suppurative Appendicitis
Brief Title: Fast Track Appendectomy for Suppurative Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13-0660
Record Dates: First submitted 2014-05-07; First posted 2014-05-14 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Suppurative Appendicitis
Keywords: Suppurative appendicitis, appendicitis, pediatric
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast track (Experimental): Patients discharged home the same day following appendectomy
  Interventions: Other: Patients discharged home the same day following appendectomy
- Admission (No Intervention): Patients are admitted to the inpatient unit following appendectomy for suppurative appendicitis and treated per the current standard of care.

INTERVENTIONS:
Other: Patients discharged home the same day following appendectomy — Patients are discharged to home on the same day following appendectomy with oral antibiotics.
  Arms: Fast track

SUMMARY:
The literature has reported that fast track surgery can be safely applied to children undergoing appendectomy for acute appendicitis. There is no current evidence regarding the application of same day discharge protocol in children with intra-operative findings of suppurative appendicitis. The current standard of care for patients who present with intra-operative findings of suppurative appendicitis includes post-operative admission and treatment with intravenous antibiotics. Patients are discharged home once they have met the following discharge criteria: temperature less than 38.5 degrees Celsius, pain control with oral pain medication, and tolerating a liquid diet. Given the evidence in the literature that has shown that same day discharge of patients with acute appendicitis is safe and effective, we propose that fast track surgery protocol can be safely applied to patients with intraoperative findings of suppurative appendicitis. We hypothesize that this will result in a decreased postoperative length of stay, without an increase in 30-day complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 5-18
* Diagnosis of appendicitis and scheduled for appendectomy during the hours of 0600-1800.
* Intraoperative findings of suppurative appendicitis

Exclusion Criteria:

* Pregnancy
* Complex medical history not appropriate for same day discharge

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Chandler, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fast Track | Admission
Started | 18 | 18
Completed | 16 | 18
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fast Track | Admission | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 18 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.4) | 11.6 (3.5) | 11.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Length of Stay
Time Frame: Post anesthesia care unit arrival to discharge home, an expected average of up to 48 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Fast Track | Admission
Number analyzed (Participants) | 18 | 18
Hours | 8.2 (18.7) | 23.4 (4.2)

2. Secondary Outcome: Thirty Day Complication Rate
Description: Superficial wound infection, deep organ space infection, ileus or bowel obstruction requiring hospitalization or re-operation
Time Frame: Thirty days
Measure: Number; unit: participants
Arm/Group | Fast Track | Admission
Number analyzed (Participants) | 18 | 18
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Thirty days
Arm/Group | Fast Track | Admission
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
The small number of patients enrolled in each arm and the low number of 30-day patient follow up limit the interpretation of the current results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes